CLINICAL TRIAL: NCT02349737
Title: Use of Bioelectrical Impedance Analysis in the Nutritional Assessment of Patients With CHF Equipped With Implantable Cardioverter Defibrillators
Brief Title: Evaluation of Interference Between Bioelectrical Impedance Analysis and Implantable Cardioverter Defibrillators
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Philippe Meyer, MD, University Hospital, Geneva
Other Study IDs: Quality control study
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Electromagnetic Interference
Keywords: Bioelectrical Impedance Analysis; Body composition; ICD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Electromagnetic Interference
  Interventions: Other: Exposure to BIA interference with the ICD

INTERVENTIONS:
Other: Exposure to BIA interference with the ICD — Exposure to BIA interference with the ICD
  Other Names: Study group

SUMMARY:
Evaluation of electromagnetic interference between Bioelectrical Impedance Analysis (BIA) and implantable cardioverter defibrillators (ICDs).

DETAILED DESCRIPTION:
Electrograms of ICDs will be analyzed during wireless telemetry and during body composition measurement using BIA. ICD therapy will have been temporarily inactivated before the measurement to avoid inappropriate shocks, and the sensitivity level of the ICD will be set to maximum. Body composition will be measured at three frequencies (5 khz, 50 khz and 100 khz).

Interference will be assessed by the presence of visible artefacts on the real-time electrogram, with ICD marker annotations showing atrial and/or ventricular sensed episodes. The outcome measure will be the number and proportion of patients who have electromagnetic interferences of the ICD when BIA is done.

The procedure will take approximately 5-10minutes, with reprogramming of the device at the end of the test. No further follow-up in the context of the study will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Implantation with a wireless-enabled ICD

Exclusion Criteria:

* Age <18yrs
* Inability to sign an informed consent
* Pacemaker dependancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ICD.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who have electromagnetic interference of the ICD when exposed to BIA. | 5-10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Buch E, Bradfield J, Larson T, Horwich T. Effect of bioimpedance body composition analysis on function of implanted cardiac devices. Pacing Clin Electrophysiol. 2012 Jun;35(6):681-4. doi: 10.1111/j.1540-8159.2012.03377.x. Epub 2012 Mar 27. PMID 22452409
- [Derived] Meyer P, Makhlouf AM, Mondouagne Engkolo LP, Trentaz F, Thibault R, Pichard C, Burri H. Safety of Bioelectrical Impedance Analysis in Patients Equipped With Implantable Cardioverter Defibrillators. JPEN J Parenter Enteral Nutr. 2017 Aug;41(6):981-985. doi: 10.1177/0148607116633823. Epub 2016 Feb 22. PMID 26903305